CLINICAL TRIAL: NCT02198118
Title: Domiciliary Physiotherapy During Breast Cancer Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Helio Carrara, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCT01940107; USP-HCarrara (Other: University of São Paulo)
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Shoulder Pain
Keywords: breast cancer; physiotherapy; radiotherapy
MeSH Terms: conditions — Shoulder Pain; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Control group (CG) subjected only to evaluations and to no exercises.
- Study Group (Experimental): Study group (SG) instructed to perform domiciliary exercises for the upper limbs
  Interventions: Other: Domiciliary exercises for the upper limbs

INTERVENTIONS:
Other: Domiciliary exercises for the upper limbs — Study group (SG) instructed to perform domiciliary exercises for the upper limbs.
  Arms: Study Group

SUMMARY:
Background: Breast cancer is the most common type of cancer among women. Its treatment, including radiotherapy (RT), can cause potential complications to be treated by the physiotherapy. Objective: To evaluate the effect of domiciliary physiotherapy on the upper limb applied during the period of radiotherapy in women submitted to surgical and radiotherapy for breast cancer. Study design: This is a prospective randomized controlled clinical trial. Methods: Thirty six volunteers were recruited from November 2009 to March 2012 and they were appraised at three different times: pre-RT, post-RT and 2 months after the end of RT. The parameters evaluated were: shoulder range of movement (ROM) and arm circumference. They were divided into two groups: CG) control group, submitted only to the assessments and SG) study group, submitted to domiciliary physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Having been diagnosed with unilateral breast cancer and having been submitted to surgical and radiation treatment as part of the treatment for breast cancer, according to the therapeutic protocol of the unit

Exclusion Criteria:

- Patients with neurological or orthopedic diseases that could impair the movements of the upper limbs, bilateral breast cancer, previous thoracic radiotherapy, and the presence of distant metastasis.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gain in range of movement measured in degrees | Three months
  The volunteers were evaluated at three distinct times: pre-RT (first evaluation), post-RT (second evaluation) and 2 months after the end of RT (third evaluation). The following parameters were evaluated: ROM of shoulder joint and upper limb perimetry. To assess shoulder ROM, the movements of flexion, extension, abduction, adduction, internal rotation and external rotation were measured, with each movement being performed by subjects. The volunteers were randomly divided into 2 groups: a control group (CG) subjected only to evaluations and to no exercise, and a study group (SG) instructed to perform domiciliary exercises for the upper limbs. The plan randomization was performed by a computer program that generated a list with the allotment of cases to the two groups. The allocation was randomized, but not concealed.

SECONDARY OUTCOMES:
Improvement of lymphedema measured in centimeters | Three months
  Lymphedema was evaluated during the period of the study through perimetry measurements that were made at 6 different points: point A -metacarpophalangeal joint of the 2nd, 3rd, 4th and 5th fingers; point B - an imaginary line passing through the metacarpophalangeal joint of the thumb; point C - 10 cm below the olecranon; point D - 6 cm below the olecranon; point E - 6 cm above the olecranon, and point F - 10 cm above the olecranon 20. The volunteer should be sitting, with her arm resting on her thigh and the forearm supinated. The measurements were bilateral and carried out by the same observer.

CONTACTS AND LOCATIONS:
Overall Officials: Nara FB Leal, Master, Study Chair — University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Leal NF, Oliveira HF, Carrara HH. Supervised physical therapy in women treated with radiotherapy for breast cancer. Rev Lat Am Enfermagem. 2016 Aug 15;24:e2755. doi: 10.1590/1518-8345.0702.2755. PMID 27533265